CLINICAL TRIAL: NCT04007601
Title: Neurostimulation In Adult Survivors of Childhood Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NEUROSTIM; R01CA239630 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Neurocognitive impairment; Executive dysfunction; Survivorship
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Active Comparator): Remotely delivered active tDCS + cognitive training
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator): Remotely delivered sham tDCS + cognitive training
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Participants will receive active 1mA direct current stimulation over the left dorsolateral prefrontal cortex for 20 minutes. Cognitive training: Participants will complete 20 minutes of online cognitive training via Lumosity two days per week for a 6-month intervention period.
  Arms: Active tDCS
Device: Sham tDCS — Participants will receive sham (no direct current) stimulation over the left dorsolateral prefrontal cortex for 20 minutes. Cognitive training: Participants will complete 20 minutes of online cognitive training via Lumosity two days per week for a 6-month intervention period.
  Arms: Sham tDCS

SUMMARY:
Long-term survivors of ALL are at-risk for neurocognitive impairment, particularly in the area of executive functioning. Relatively limited research has focused on interventions for improving neurocognitive outcomes in long-term survivors of ALL. A promising technique for cognitive enhancement is Transcranial Direct Current Stimulation (tDCS) which differs from conventional cognitive remediation approaches in that it directly stimulates specific brain regions responsible for cognitive processes and activates functional networks similar to those activated during cognitive training.

Primary Objective

To evaluate the efficacy of home-based transcranial direct current stimulation (tDCS) paired with remote cognitive training on direct testing of executive function in survivors of ALL.

Secondary Objectives

* To evaluate the efficacy of home-based transcranial direct current stimulation (tDCS) paired with remote cognitive training on patient-reported symptoms of executive dysfunction in survivors of ALL.
* To examine the effects of home-based tDCS paired with remote cognitive training on patterns of regional brain activation as measured by functional magnetic resonance imaging.
* To examine the effects of home-based tDCS paired with remote cognitive training on white matter integrity and structure as measured by diffusion tensor imaging.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive 1 mA direct current stimulation over the left dorsolateral prefrontal cortex or placebo/sham for 20 minutes. All participants will receive home-based computerized cognitive training. Participants will complete tDCS paired with cognitive training 2 times per week for 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for acute lymphoblastic leukemia (ALL) at SJCRH < 21 years at diagnosis
* Enrolled on St. Jude Lifetime Cohort Study
* ≥ 5 years post-diagnosis of ALL
* ≥ 2 years post-treatment completion deemed to impact the central nervous system.
* Currently between 18 and 39 years of age
* English language proficiency
* Executive dysfunction defined as having an age-adjusted standard score <16th percentile on Trail Making Test Part B, Controlled Oral Word association Test, or Digit Span Backward
* Patient-reported executive dysfunction defined as a standard score >84th percentile on the Childhood Cancer Survivor Study Neurocognitive Questionnaire or the Behavior Rating Scale of Executive Function

Exclusion Criteria:

* Full scale intelligence score <80
* Currently taking medication intended to treat neurocognitive impairment (e.g. stimulants)
* Participated in a past trial of neurostimulation
* Female who is pregnant or breastfeeding
* History of seizures within the past year
* Implanted medical devices or metal in the head
* History of head injury or a neurodevelopmental disorder (i.e. genetic disorder, hypoxic-ischemic encephalopathy) associated with neurocognitive impairment and unrelated to cancer treatment
* Currently receiving cancer directed therapy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Direct Testing of Executive Function: Change in Working Memory from baseline to 6 months | Baseline & 6-month follow-up
  Digit Span Backward: Digit Span Backward (DSB), from the Digit Span subtest on the WAIS-IV, is a measure of working memory. The number of digits recalled in the longest span is converted to a standard z-score using age-based norms (Mean=0, SD=1).
Direct Testing of Executive Function: Change in Cognitive Flexibility in baseline to 6 months | Baseline & 6-month follow-up
  Trail Making Test Part B (Trails B): This is a timed task that requires a participant to shift his/her attention adaptively and flexibly. Age-based standardized z-scores are calculated (Mean=0, SD=1).
Direct Testing of Executive Function: Change in Verbal Fluency from baseline to 6 months | Baseline & 6-month follow-up
  Controlled Oral Word Association (COWA): This is a task of cognitive/verbal fluency that measures spontaneous production of words beginning with a designated letter or category. Age-based standardized z-scores are calculated (Mean=0, SD=1).

SECONDARY OUTCOMES:
Change in Patient-Reported Symptoms of Executive Functioning from baseline to 6 months | Baseline and 6-month follow-up
  Patient reported symptoms of executive dysfunction will be evaluated via the Childhood Cancer Survivor Study Neurocognitive Questionnaire (CCSS-NCQ). The CCSS-NCQ is a 32-item questionnaire evaluating 4 domains of executive function. Z-scores (M=0, SD=1) are calculated using sibling data from the Childhood Cancer Survivor Study.
Change in Patient-Reported Symptoms of Executive Functioning from baseline to 6 months | Baseline and 6-month follow-up
  Patient reported symptoms of executive dysfunction will be evaluated via the Behavior Rating Inventory for Executive Function - Adult Version (BRIEF-A). The BRIEF-A is a 75-item measure of executive function that provides age- and sex-specific national normative data for nine domains of executive function (T-Score, M=50, SD=10).
Change in Brain Connectivity from baseline to 6 months | Baseline and 6-month follow-up
  White connectivity will be measured via diffusion tensor imaging and resting state fMRI (rsFMRI). The cortex will be parcellated into anatomical regions based on the high-resolution T1-weighted imaging using the FreeSurfer software (http://surfer.nmr.mgh.harvard.edu/). Probabilistic fiber tracking will be performed for individual seed points within the gray matter/white matter surface for each parcellated cortical region to evaluate strength of the connectivity between each individual region and every other region. The current project will focus analyses on the frontostriatal connections from the DLPFC to the striatum. rsfMRI data will be used to construct functional connectomes for each participant at each time point. We will measure several common connectome properties including global and local efficiency. Connectome modularity, degree distribution, and hub characteristics will also be measured.
Change in Regional Brian Activation from baseline to 6 months | Baseline and 6-month follow-up
  Regional brain activation will be assessed using an N-Back Task. This task requires a participant to respond to a presented stimulus only when it is the same as one presented on a trial at a predetermined number prior to the current trial. For this study, we plan to use 1-back and 2-back trials. Improved efficiency will be defined as reduced activation in dorsolateral prefrontal cortex during performance on the N-Back task during the fMRI. Using Statistical Parametric Mapping software (SPM12, Wellcome Trust Centre for Neuroimaging, London), contrast-images from the fixed-effect analysis in each subject will be used for second level random-effect analysis to create group activation maps. These contrasts include pre- v. post-intervention imaging during the N-back task. Participants assigned to active stimulation will then be contrasted to those assigned to sham stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols